CLINICAL TRIAL: NCT06427902
Title: Salivary Biomarkers of Gingival Inflammation Are Associated With Depression
Brief Title: Inflammatory Biomarkers in Saliva at Depression
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, DUYGU ILHAN, Asst. Prof, Medipol University
Other Study IDs: Depression
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Gingivitis; Depression; Inflammation; Inflammatory Response
MeSH Terms: conditions — Gingivitis; Depression; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- depression with gingivitis (DG) group: The diagnosis of depressive disorder was established using the Structured Clinical Interviews for Axis I Disorders (SCID) criteria of the Diagnostic and Statistical Manual of Mental Disorders.
  the gingivitis group was determined by the criteria of pocket depth of 3 mm or less.
  Interventions: Other: Periodontal clinical measurements, Saliva sampling
- depression with periodontally healthy (DPH) patients: The diagnosis of depressive disorder was established using the Structured Clinical Interviews for Axis I Disorders (SCID) criteria of the Diagnostic and Statistical Manual of Mental Disorders.
  Interventions: Other: Periodontal clinical measurements, Saliva sampling
- systemically and periodontally healthy (SPH) individuals: This group contists of individuals who are systemically and periodontally healthy
  Interventions: Other: Periodontal clinical measurements, Saliva sampling

INTERVENTIONS:
Other: Periodontal clinical measurements, Saliva sampling — Clinical periodontal indices; Probing depth, Clinical attachment level, bleeding on probing, gingival index, and plaque

SUMMARY:
The goal of this observational study is to evaluate the inflammatory saliva biomarkers in depression and gingivitis.

The main question will be ; Will there be an increase at salivary biomarkers with depression patients and is it associated with gingivitis?

DETAILED DESCRIPTION:
Background: The neuroimmune regulation disorder in depression patients causes the progression of inflammatory periodontal disease. The present study was to evaluate the periodontal health status and the levels of Triggering receptor expressed on myeloid cells 1 (TREM-1), peptidoglycan recognition protein 1 (PGLYRP1) and interleukin-1 beta (IL-1β) in individuals diagnosed with depression and to compare these findings with those of systemically healthy individuals.

Methods: Forty-two depression patients were classified in two groups: depression with gingivitis (DG) and depression with periodontally healthy (DPH) patients. Additionally, 23 systemically and periodontally healthy (SPH) individuals were enrolled to the study. Periodontal parameters were recorded. Saliva samples were collected and salivary levels of TREM-1, PGLYRP1, IL-1β were measured using Enzyme-linked Immunosorbent Assay (ELISA) kits.

depression regardless of periodontal status.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were moderate in severity according to the test result, who had not started drug therapy yet and who had not received antidepressant medication in the last 12 months

Exclusion Criteria: Patients with

* psychotic disorders
* autism spectrum disorders
* other anxiety disorders
* bipolar disorder
* mental any organic mental disorder and
* smokers, substance users

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was carried out on 65 participants in total, including 42 individuals who applied to Aydın State Hospital Psychiatry Outpatient Clinic, diagnosed with depressive disorder, were classified in 2 different groups; depression with gingivitis (DG), depression with periodontally healthy (DPH) patients and 23 systemically and periodontally healthy (SPH) individuals who applied to Adnan Menderes University Faculty of Dentistry.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
SalivaryTREM-1 | 06-09 2019
  Both, soluble and membrane-bound TREM-1, are detected by the TREM-1 ELISA.
Salivary PGLYRP1 | 06-09 2019
  Both, soluble and membrane-bound PGLYRP1 are detected by the PGLYRP1 ELISA.
Salivary IL-1β | 06-09 2019
  Both, soluble and membrane-bound IL-1β detected by the IL-1β ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Duygu Ilhan, Istanbul, Select State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided